CLINICAL TRIAL: NCT02491385
Title: Effect of Thoracic Epidural Analgesia on Bowel Function Recovery in Major Upper Abdominal Surgeries
Brief Title: Thoracic Epidural for Postoperative Ileus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyun Joo Ahn, Associate professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-12-129
Record Dates: First submitted 2015-06-30; First posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Ileus
Keywords: Thoracic epidural analgesia; bowel function recovery
MeSH Terms: conditions — Ileus | interventions — Tea; Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TEA (Experimental): thoracic epidural analgesia group
  Interventions: Procedure: thoracic epidural analgesia
- iv-PCA (Active Comparator): intravenous patient controlled analgesia group
  Interventions: Drug: iv-PCA

INTERVENTIONS:
Procedure: thoracic epidural analgesia — In a sitting position, an 18-gauge Tuohy needle is introduced at T6-7 or T7-8 intervertebral space using a paramedian approach. An epidural catheter is advanced 5 cm beyond the tip of the needle and secured with a sterile dressing. For TEA regimen, hydromorphone (8 mcg/ml) was added to 0.15% ropivacaine. TEA setting was bolus/lock out time/basal, 3 ml/15 min/5 ml.
  Arms: TEA
Drug: iv-PCA — iv-PCA setting was fentanyl 20 mcg/ml, bolus/lock out time/basal, 0.5 ml/15 min/0.5 ml.
  Arms: iv-PCA

SUMMARY:
The investigators try to find whether thoracic epidural analgesia (TEA) shortens the first gas-out time compared to iv-PCA and promotes earlier discharge after major upper abdominal surgery.

DETAILED DESCRIPTION:
Postoperative ileus (POI) is a prolonged inhibition of coordinated bowel activity after surgery. Half of patients undergoing major abdominal surgery experience POI making it one of the limiting factors for early recovery.

The pathogenesis of POI is multifactorial, and includes neurogenic, inflammatory and pharmacological mechanisms. Thoracic epidural analgesia (TEA) can induce sympathetic block, attenuate inflammatory reaction and limit use of systemic opioids. In addition, sympatholysis induced by TEA can improve microcirculation of bowels and parasympathetic activation can increase gastrointestinal motility.

However, studies comparing TEA and iv-PCA on POI are rare in major upper abdominal surgeries. This study, therefore, compares TEA and iv-PCA in terms of bowel function recovery as a primary endpoint in major upper abdominal surgeries. Secondary endpoints are side effects and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists' (ASA) physical statusⅠ-Ⅲ

Exclusion Criteria:

* ASA status of Ⅳ, or more
* Body mass index 30 kg.m2-1 or more
* Severe renal, hepatic, or neurologic diseases
* Opioid or systemic analgesic preoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
gas out time | from operation to post operative 10 days

SECONDARY OUTCOMES:
voiding time | from operation to post operative 10 days
numeric rating scale for pain | from operation to post operative 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Joo Ahn, Professor, Principal Investigator — Department of Anesthesiology and Pain Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung medical center, Seoul, South Korea